CLINICAL TRIAL: NCT02570555
Title: Strabismus Surgery and Driving Ability
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5503
Record Dates: First submitted 2013-02-12; First posted 2015-10-07 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Strabismus; Esotropia; Exotropia
Keywords: driving
MeSH Terms: conditions — Strabismus; Esotropia; Exotropia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The strabismus impacts binocular visual acuity and stereoscopy. Thus, driving capacities of patients with strabismus may be reduced. The goal of this work is to study the possible amelioration of driving ability after strabismus surgery and to compare the driving capacities of patients with strabismus to a normal population; Patients will be tested before and after strabismus surgery using a driving simulator, binocular visual field and binocular visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Strabismus
* Age > 18 yrs old
* Driving license

Exclusion Criteria:

* Inability to driving under French law

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with strabismus tested before and after the eye surgery Control patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of strabismus surgery on driving ability by using a Performance score (number of errors, braking velocity, speed variations of the vehicle position). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Sauer, MDPHD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Sevice d'ophtalmologie Les hôpitaux Universitaires de Strasbourg, Strasbourg, France